CLINICAL TRIAL: NCT02002078
Title: High Doses of Methylprednisolone in the Management of Caustic Esophageal Burns in Children
Brief Title: Caustic Esophageal Burns in Children and High Doses of Methylprednisolone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Usta, DR, Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: ClinicalTrials.gov
Record Dates: First submitted 2013-11-22; First posted 2013-12-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: Esophageal Diseases
Keywords: caustic; corticosteroid therapy; stricture; children
MeSH Terms: conditions — Esophageal Diseases; Constriction, Pathologic | interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methylprednisolone, caustic burns (No Intervention)
  Interventions: Drug: methylprednisolon

INTERVENTIONS:
Drug: methylprednisolon

SUMMARY:
Corrosive substance ingestion in childhood is a public health issue in developing countries and several management protocols were proposed to prevent esophageal strictures. The role of corticosteroids in preventing corrosive-induced strictures is controversial. The investigators' aim is to study the influence of high doses of corticosteroids to prevent esophageal strictures.

ELIGIBILITY:
Inclusion Criteria:

-Corrosive substance ingested children with grade IIb esophageal burn

Exclusion Criteria:

* Caustic substance ingested chldren grade I, IIa and grade III esophageal burns
* Caustic subtance ingested children with signs of perforation, mediastinitis, peritonitis, sespis
* Caustic substance ingested children with any chronic disease

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of stricture development in children with caustic esophageal burns after high doses of methylprednisolone | three years
  stricture development was evaluated with endoscopic examination and upper gastrointestinal system series with barium swallow

REFERENCES:
- [Derived] Usta M, Erkan T, Cokugras FC, Urganci N, Onal Z, Gulcan M, Kutlu T. High doses of methylprednisolone in the management of caustic esophageal burns. Pediatrics. 2014 Jun;133(6):E1518-24. doi: 10.1542/peds.2013-3331. PMID 24864182